CLINICAL TRIAL: NCT03889704
Title: Neuromuscular Electrical Stimulation for Jaw-closing Dystonia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic
Sponsor: Edward Burton (Other)
Responsible Party: Sponsor-Investigator, Edward Burton, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY18120054
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Muscle Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neuromuscular electrical stimulation (Experimental): The Omnistim® FX² is a neuromuscular stimulation device that provides patterned electrical neuromuscular stimulation (PENS) via cutaneous electrodes placed over relevant musculature. It will be applied for 20 minutes per session. For each patient, there will be 2 sessions per week, spaced 3 to 4 days apart. Each patient will participate in 16 sessions over the 8 weeks of the study. There will be 6 patients total.
  Interventions: Device: Omnistim® FX²

INTERVENTIONS:
Device: Omnistim® FX² — The Omnistim® FX² is a neuromuscular stimulation device that provides patterned electrical neuromuscular stimulation (PENS) via cutaneous electrodes placed over relevant musculature. The device mimics physiologic patterns of neuron firing.

SUMMARY:
6 patients with jaw-closing dystonia will be treated with neuromuscular electrical stimulation over 8 weeks. The distance the mouth can be opened voluntarily and the oro-mandibular dystonia questionnaire (OMDQ-25) will be employed to determine whether there is any objective change in jaw opening or evidence of functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* Jaw-closing dystonia, which may be primary or secondary to a neurodegenerative disease or medications.
* Unable to voluntarily open jaw fully on examination.
* Evidence of functional impairment resulting from dystonia including inability to completely open the jaw during speaking or eating to such an extent that it interferes with these tasks.
* Patient interested in participating, and willing to attend multiple treatment sessions in the neurology clinic.

Exclusion Criteria:

* Presence of a cardiac pacemaker, implanted defibrillator, or other implanted electronic device.
* Inability to provide consent (either by the patient, spouse, or an identified power of attorney).
* Age under 18 years.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Burton, MD, DPhil, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neuromuscular Electrical Stimulation
Started | 2
Completed | 1
Not Completed | 1
Not completed — Study terminated due to pandemic | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 72 [69 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Jaw Opening
Description: Measured via tongue depressor quantity, which is the number of stacked tongue depressors the patient is able to safely fit between his or her incisors.
Time Frame: Change from before starting first treatment to after completing last treatment, usually completed over 8 weeks.
Measure: Mean (Full Range); unit: tongue depressors
Arm/Group | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 2
tongue depressors | 3 [3 to 3]

2. Primary Outcome: Jaw Opening
Description: as for outcome 1
Time Frame: Average change from before to after each 20-minute treatment session.
Measure: Mean (Full Range); unit: Tongue depressors
Arm/Group | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 2
Tongue depressors | 0.0813 [0.0625 to 0.1]

3. Primary Outcome: Oromandibular Dystonia Questionnaire
Description: Questionnaire that assesses quality of life in oromandibular dystonia patients. There are 25 questions total, and each question may be answered as never, seldom, sometimes, often, always. Minimum score is 0, maximum score is 100. A higher score indicates worse quality of life.
Time Frame: Change from before the first treatment to after the last treatment, usually over 8 weeks.
Measure: Mean (Full Range); unit: score on a scale (OMDQ25)
Arm/Group | Neuromuscular Electrical Stimulation
Number analyzed (Participants) | 2
score on a scale (OMDQ25) | -21 [-29 to -13]

ADVERSE EVENTS:
Time Frame: During participation in the study (16 sessions)
Description: Patients were evaluated for any adverse effects during or after treatment at each session, and before treatment for AEs arising after the previous treatment.
Arm/Group | Neuromuscular Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Owing to pandemic restrictions, the study only recruited 2 patients prior to termination and only 1 completed all sessions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03889704/Prot_000.pdf